CLINICAL TRIAL: NCT04271995
Title: A Diagnostic Accuracy Study Evaluating Point of Care Gastric Lipase Enhanced pH Test Strip to Confirm Correct Nasogastric Tube Position in Newborn Infant
Brief Title: Gastric Lipase Enhanced Nasogastric Tube Study in Neonates
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19QC5444
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Neonatal Disorder
Keywords: nasogastric tube; gastric lipase
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The newborn infants who are sick and those who are born prior to due date (preterm) are admitted to the neonatal unit. These babies are unable to feed through their mouth, so a special tube is passed through their nose to the stomach, nasogastric (NG) tube) to provide milk feeds. The bedside nurse inserts the tube and then aspirate some of the fluid from the stomach. As the stomach normally produce acid, these aspirate is then tested on a colour coded paper strip to check if the fluid is acidic. However, on many occasions this test is not very clear. This could be due to misplacement of the tube or the stomach in a newborn not being able to produce enough acid. This then leads to re-siting of another tube and following the same procedure. Sometimes the clinical team may like to do an X Ray to check the position of the tube resulting in unnecessary exposure to radiation. The study will use a special chemical added to the currently existing paper test strip which the investigators believe will enhance the capability of detecting the correct position of the NG tube. This idea has been tested in adults and found to have increased the sensitivity of the test strip significantly. Based on the adult study the study will require to test 233 babies to see if this increases the sensitivity of correct NG tube placement. Parents of all babies who requires an NG tube for milk feeds will be approached and after appropriate consent could be recruited to the study. Babies who are clinically very unstable, moribund and those with diagnosis of bowel obstruction will be excluded from the study.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objective:

• To determine the sensitivity of the chemical (tributyrin) impregnated pH test strip in comparison to the routine pH test strip to increase the sensitivity of detection of correct positioning of the nasogastric tube

Secondary objectives:

* To measure the number of nasogastric tube re-insertion attempts that could be avoided if the tributyrin impregnated pH test strip was used instead of the standard pH test strip
* To determine the number of chest radiographs which could be avoided if the tributyrin impregnated pH test strip was used instead of the standard pH test strip
* To carry out human factors assessment of perceived usability, trust and acceptance of the lipase-based pH test strip

STUDY DESIGN Prospective point of care diagnostic accuracy study

Primary outcome

• Sensitivity of proposed test in determining correct nasogastric (NG) tube position

Secondary outcomes

* Number of chest x rays performed
* Time to confirm tube placement
* Number of nasogastric tube attempts to get the correct pH
* Assessment of human factors - Perceived usability, trust and acceptance from professionals' perspective

Subject selection and setting

Participants will be recruited from Imperial College Healthcare NHS Trust from the neonatal units at both the Queen Charlotte's and Chelsea and St. Mary's hospital sites. Eligible participants will be identified by the clinical team and recruited by a member of the research team.

The vast majority of admitted infants will require nasogastric tube insertion as part of their clinical management such as preterm infants, sick term infants with hypoxic- ischaemic encephalopathy and meconium aspiration syndrome as well as admitted infants for hypoglycaemia and jaundice management.

Study method

The clinical trial will be a diagnostic accuracy study of two diagnostic tests and will be reported in accordance with the Standards for reporting diagnostic accuracy studies (STARD) guidelines. The index tests will be (i) the novel tributyrin impregnated pH test strip and (ii) standard pH test strip. The reference test used for comparison will be chest x-ray performed earlier or later but with the same nasogastric tube in situ; or where this is not required 'trial by use' (any chest x-rays undertaken would be decided and authorised by the participant's clinical team who are clearly separated from the research team. Undergoing a chest x-ray does not from part of screening for the study and is not a requirement of the study protocol).

Ingenza novel lipase/pH test strip

The test detects the organic acid released from tributyrin, a chemical ester impregnated onto pH paper by the action of human gastric lipase that is stable in gastric juice and resistant towards antacid medications, as well as unlikely to migrate. Ingenza have impregnated enteral pH indicator strips that are in current clinical use with emulsion formulations of tributyrin, protected by intellectual property as human gastric lipase substrates. Therefore, the novel test strips will provide a positive result in the presence of an acidic environment (pH less than or equal to 5.5) or gastric lipase.

Index testing

After the tube insertion, the carer will aspirate the tube to obtain a sample of gastric fluid. This will be done immediately following insertion or as part of daily position confirmation that is routinely performed prior to initiation of nasogastric feeding. The aspirate will be used by the healthcare professional, as part of routine care and the remaining sample passed to a member of the research team. The healthcare professional will test the aspirate routinely and make their decision based on the current standard pH strip test. The remaining sample will be used by the research nurse blinded to the standard test, to wet the gastric lipase enhanced pH test strip. The research nurse will then independently assess the results of the study test paper at two minutes. Digital photographs of both the routine and the study test papers will be assessed independently by member of the study team to verify the findings. The healthcare professional will be blinded to the results of the proposed test strip. The research nurse will record the results of the standard test strip only after documenting the result of the proposed test.

For standard pH strips a pH of ≤5.5 will indicate correct tube placement and >5.5 indicates incorrect nasogastric tube position. For the gastric lipase enhanced pH strip test a positive result will be determined according to the manufacturer's recommendations.

INCLUSION CRITERIA

All infants (preterm and term) who require the insertion of nasogastric tubes for supplementary enteral feeding as part of their routine clinical management

EXCLUSION CRITERIA

Clinically unstable, critically ill infants Infants undergoing palliative care Infants with bowel conditions such as necrotising enterocolitis, bowel obstruction

ELIGIBILITY:
Inclusion Criteria:

* All infants (preterm and term) who require the insertion of nasogastric tubes for supplementary enteral feeding as part of their routine clinical management

Exclusion Criteria:

* Clinically unstable, critically ill infants
* Infants undergoing palliative care
* Infants with bowel conditions such as necrotising enterocolitis, bowel obstruction

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants admitted to the neonatal unit requiring insertion of nasogastric tube
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of standard and ingenza pH strips | 6 months
  Where test sensitivity is defined as the proportion of pH readings that are equal to or below (<=) a certain cut-off when aspirates are obtained from tubes placed inside the stomach. Stomach placements are confirmed either by chest x-rays, or in its absence, by clinical observations).

SECONDARY OUTCOMES:
Number of chest x rays performed | 6 months
  Number of chest X Rays performed to confirm nasogastric tube position after insertion and failure of detection of position using currently available pH measurement strips
Time to confirm tube placement | 6 months
  Total time in minutes to confirm nasogastric tube position
Number of nasogastric tube attempts to get the correct pH | 6 months
  Number of nasogastric tube attempts to get the correct pH
Specificity of standard and ingenza pH strips | 6 months
  Where test specificity is defined as the proportion of pH readings that are greater than (>) a certain cut-off when aspirates are obtained from tubes placed outside the stomach. Non-stomach placements are confirmed by chest x-rays or through reported adverse events.
pH readings obtained by standard and ingenza strips under all cut-offs | 6 months
  pH readings obtained by standard and ingenza strips under all cut-offs

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom